CLINICAL TRIAL: NCT05675176
Title: Antegrade Observational Comparative Study for the Intravesical Instillation Therapy of Bacillus Calmette Guerin With the Use of Different Types of Urinary Catheters in Patients With Urinary Bladder Cancer
Status: Completed | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Bellos Themistoklis, Doctor of Medicine, National and Kapodistrian University of Athens
Other Study IDs: 15306/26-7-22
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Non-muscle-invasive Bladder Cancer
Keywords: bladder cancer; intravesical instillation; complications; BCG; hematuria; fever; LUTS; Tuberculosis
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms; Hematuria; Fever; Tuberculosis | interventions — Administration, Intravesical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients with non muscle invasive bladder cancer undergoing intravesical instillation with the use of self lubricated silicon tiemann 10 fr urinary catheter.
  Interventions: Drug: BCG
- Group 2: Patients with non muscle invasive bladder cancer undergoing intravesical instillation with the use of straight tipped latex foley 14 fr urinary catheter
  Interventions: Drug: BCG

INTERVENTIONS:
Drug: BCG — Intravesical Instillation
  Other Names: Intravesical Instillation

SUMMARY:
The study compares the complications caused after the BCG intravesical instillation in patients treated for non invasive bladder cancer.The patients are divided into two groups one receiving IVI (intravesical Instillations) with the use of latex catheter while in the other silicone catheter is used.The two groups are compared in terms of fever, hematuria, LUTS and other complications following IVI.

DETAILED DESCRIPTION:
Bladder cancer is the 9th most common diagnosed cancer according to 2021 statistics (4). It can be divided into muscle invasive (MIBC) and non muscle invasive bladder cancer (NMIBC) , based on the biopsy result after transurethral resection of the bladder tumor.In this research we will abide ourselves to the non muscle invasive bladder cancer.After the transurethral resection of bladder cancer, further management of this disease includes the intravesical instillation of chemotherapy or immunotherapeutic drugs.

The most commonly used drugs in our clinic is epirubicin and Bacillus Calmette Guerrin (BCG) for intravesical instillations.This research will focus on the use of intravesical instillations of BCG .Intravesical instillations of BCG are performed in patients with pTa/High Grade (HG), pT1/Low Grade(LG), pT1/HG and Carcinoma in Situ(CIS) tumors , while epirubicin is used in tumors pTa/LG.

The most common complications after intravesical instillation of BCG are either systemic (mycotic aneyrysms , tuberculosis, hepatitis, arthritis , spondylitis or ev enencephalitis) or are related to the urogenital system (cystitis, prostatitis which can be either tuberculous or bacterial, balanitis or tuberculous epididymitis) (3). The most common complications of the urinary system after the intravesical BCG instillation can appear as a combination of the lower urinary tract symptoms (LUTS) , macroscopic hematuria and fever (4).

There are researches that prove the superiority of silicon catheters for long term catheterization in terms of reduced urethral inflammation and consequently reduced LUTS (1,2). However, there is also an article that claims that latex urinary catheters that are coated with noble metals cause minimal LUTS compared with silicone catheters when used for short term catheterization (3). Nevertheless, there is not a comparative antegrade study for the use of different type of catheters for the intravesical instillation of BCG that proves the superiority of one catheter type over the other.

Purpose of this study The purpose of this study is the comparison of the symptoms arising from the use of two different types of urinary catheters (latex or silicon tiemann) during the intravesical instillation of BCG and the possible display of superiority of one of those catheter types.

Material and Methods This study is an antegrade comparative cohort study. In this are included patients of all age and genders. The patients were diagnosed with non muscle invasive bladder cancer after the transurethral resection of the bladder tumor and are undergoing intravesical BCG instillations after they get their biopsy results.They undergo either 6 weekly intravesical instillations in de novo diagnosed cancer or in 3 weekly instillations during the follow-up based on our clinic's protocol. The intravesical therapy begins 2-4 weeks after the surgery , since the patients has a negative urine culture. Another important condition is that the patient does not have macroscopic hematuria ,does not have fever or does not bleed during the catheter insertion.

The intravesical instillation is performed in the outpatient department of the 2nd University Urology Clinic in Sismanogleio Hospital ,Athens, Greece by three urologist J.M. ,T.B. and S.K.. Those three physicians use aseptic and non traumatic technique during the intravesical instillations (IVIs). For the IVIs either self lubricated silicon tiemann 10 fr urinary catheter or straight tipped latex foley 14 fr urinary catheter was used. The catheterization was done with the use of 2% xylocaine jelly in the urethra.The catheter was advanced slowly while the intravesical instillation was done slowly in a rate so that it was completed in 20-30 s.This technique was used by all the physicians.

The preparation and dilution of the drug used for the IVIs was done by the same trained nurses, under the same conditions for each case and is instilled as soon as it is ready.Before every insillation the physician asks the patient if he has symptoms since the previous instillation such as macroscopic hematuria, fever or LUTS. In case that one of those symptoms exists then the instillation is not performed.In case of hematuria ,instillation is postponed until this symptom disappears.In case of persisting LUTS until the the next instillation the patient receives antibiotic regimen based on urinary culture and continues with the instillation when the culture is negative. In case of fever above 38 celsius the patient undergoes an empiric antibiotic regimen with quinolones. If fever persists over 48 hours then the patient is reffered to an internist with subspecialisation in infectious medicine to exlude the possibility of systemic or urogenital tuberculous complication. The intravesical instillation regimen continues when the patient has no longer fever.

ELIGIBILITY:
Inclusion Criteria:

* BCG intravesical instillation for non muscle invasive bladder cancer

Exclusion Criteria:

* Positive culture
* Preexisting LUTS
* Muscle invasive bladder cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with non muscle invasive bladder cancer undergoing intravesical instillation with BCG.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-04-12 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Complications | 1.5 year
  Complications in both groups- hematuria, fever, LUTS , systemic symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Themistoklis Bellos, Marathon, Attica, Greece

REFERENCES:
- [Background] Nacey JN, Tulloch AG, Ferguson AF. Catheter-induced urethritis: a comparison between latex and silicone catheters in a prospective clinical trial. Br J Urol. 1985 Jun;57(3):325-8. doi: 10.1111/j.1464-410x.1985.tb06354.x. PMID 3891005
- [Background] Stenzelius K, Persson S, Olsson UB, Stjarneblad M. Noble metal alloy-coated latex versus silicone Foley catheter in short-term catheterization: a randomized controlled study. Scand J Urol Nephrol. 2011 Sep;45(4):258-64. doi: 10.3109/00365599.2011.560007. Epub 2011 Mar 31. PMID 21452931
- [Background] Liu Y, Lu J, Huang Y, Ma L. Clinical Spectrum of Complications Induced by Intravesical Immunotherapy of Bacillus Calmette-Guerin for Bladder Cancer. J Oncol. 2019 Mar 10;2019:6230409. doi: 10.1155/2019/6230409. eCollection 2019. PMID 30984262
- [Result] Talja M, Korpela A, Jarvi K. Comparison of urethral reaction to full silicone, hydrogen-coated and siliconised latex catheters. Br J Urol. 1990 Dec;66(6):652-7. doi: 10.1111/j.1464-410x.1990.tb07203.x. PMID 2265339